CLINICAL TRIAL: NCT02096666
Title: A Multicenter, Phase 1/2, Open-Label Study Evaluating the Tolerability, Safety, Pharmacokinetics, and Efficacy of AMG 337 in Asian Subjects
Brief Title: A Phase 1/2 Study Evaluating AMG 337 in Asian Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120370
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Stomach Neoplasms
Keywords: MET Amplified Gastric/ Gastroesophageal Junction/ Esophageal Adenocarcinomas, or other solid tumors
MeSH Terms: conditions — Stomach Neoplasms | interventions — AMG 337

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: AMG 337

INTERVENTIONS:
Drug: AMG 337 — Phase 1- AMG 337 150 mg, 200mg and 300 mg orally daily. Additional 150 mg and 200 mg orally twice daily. Phase 2- AMG 337 (dose determined by Phase 1)

SUMMARY:
This is a multicenter, Phase 1/2 study. The study will evaluate the tolerability, safety and activity of AMG 337 in Asian subjects who have advanced solid tumors (Phase 1) or subjects with MET amplified tumors with a focus on gastric/gastroesophageal junction/esophageal adenocarcinoma (Phase 2).

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter, single arm, open-label study to assess the safety, efficacy and pharmacokinetics of AMG 337 in solid tumors. In the Phase 1, approximately 3 to 45 subjects enrolled in a 3+3+3 dose escalation scheme evaluating two dose levels. In the Phase 2, approximately 140 subjects will be enrolled to either Cohort 1 (subjects with MET amplified /gastroesophageal junction/esophageal (G/GEJ/E) adenocarcinoma with measurable tumor) or Cohort 2 (subjects with MET amplified solid tumors with measurable tumor and subjects with MET amplified G/GEJ/E adenocarcinoma with non-measurable tumor). All subjects will self-administer AMG 337 daily until disease progression or other protocol specified end of treatment criteria are met. Tumor assessment by RECIST 1.1 will be followed during study treatment.

Tumor tissue, biomarkers, pharmacokinetics and Patient Reported Outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to self administer daily AMG 337 as a whole capsule
* Male or female 20 years of age or over
* Phase 1: Subjects must have a pathologically confirmed, advanced solid tumor for which the subjects have received prior therapy for advanced disease, for which no standard therapy exists, or the subject refuses standard therapy.
* Phase 2: Subjects must have a pathologically confirmed, advanced G/GEJ/E adenocarcinoma (cohort 1) or other solid tumor (cohort 2) for which the subjects have received prior therapy for advanced disease, or for which no standard therapy exists, or the subject refuses standard therapy.
* Tumor MET amplified by protocol-specified centralized testing (phase 2 only).
* Phase 1: Measurable or non-measurable disease per RECIST v1.1
* Phase 2: Measurable disease per RECIST v1.1 guidelines. Cohort 2 may include subjects with advanced MET amplified G/GEJ/E adenocarcinoma with non-measurable tumor per RECIST v1.1.
* (ECOG) Performance Status of 0, 1, or 2
* Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

* Known central nervous system metastases.
* Subject is a candidate for curative surgery or definitive chemoradiation.
* Peripheral edema > grade 1.
* Subjects who have persistent gastric outlet obstruction, complete dysphagia or are dependent upon jejunostomy for feeding. Significant gastrointestinal disorder(s) that in the opinion of the Investigator may influence drug absorption.
* Currently receiving any anti-tumor treatments, or less than 14 days prior to enrollment since ending anti-tumor treatment.
* Prior treatment with small molecule inhibitors of the MET pathway.
* Other protocol defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Phase 1- Adverse events and clinical laboratory abnormalities | 17 months
  Adverse events and clinical laboratory abnormalities defined as DLTs.
Phase 2- Overall Response Rate (per RECIST v1.1) in subjects with MET amplified measurable gastric/gastroesophageal junction/esophageal adenocarcinoma (cohort 1) | 17 months
  Determine anti-tumor activity of AMG 337 in subjects with MET amplified gastric/gastroesophageal junction/esophageal adenocarcinoma (cohort 1)

SECONDARY OUTCOMES:
Phase 1- Pharmacokinetic parameters | 17 months
  Including, but not limited to, minimum (trough) concentrations, maximum concentrations (C max), the time of C max (t max), and area under the plasma concentration- time curve (AUC).
Phase 1- Other adverse events, clinical laboratory abnormalities and ECG parameters | 17 months
Phase 2- Overall Response Rate (per RECIST v1.1) in subjects with other MET amplified solid tumors (subjects with measurable disease in cohort 2) | 17 months
  Determine anti-tumor activity in AMG 337 in subjects with MET amplified solid tumors (subjects with measurable disease in cohort 2)
Phase 2- Duration of Response (cohort 1 and subjects with measurable disease at baseline in cohort 2) | 17 months
Phase 2- Time to response (cohort 1 and subjects with measurable disease at baseline in cohort 2) | 17 months
Phase 2- Progression Free Survival | 17 months
Phase 2- Overall Survival | 17 months
Phase 2- Incidence and severity of adverse events and significant laboratory abnormalities | 17 months
Phase 2- AMG 337 exposure and dose intensity | 17 months
Phase 2- Pharmacokinetic parameters | 17 months
  Including, but not limited to, minimum (trough) concentrations at pre-dose times and maximum concentrations (C max), the time of C max (t max), and area under the plasma concentration- time curve (AUC) for intensive pharmacokinetic sampling.
Phase 1- Overall Response Rate | 17 months
Phase 1- Duration of Response | 17 months
Phase 1- Time to Response | 17 months
Phase 1- Progression-Free Survival (per RECIST v1.1) | 17 months
Phase 1- Overall Survival | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Japan (4):
  - Research Site, Kashiwa-shi, Chiba
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Suntou-gun, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Yasui H, Go N, Yang H, Amore BM, Jung AS, Doi T. A Phase 1 study evaluating AMG 337 in Asian patients with advanced solid tumors. Jpn J Clin Oncol. 2017 Aug 1;47(8):772-776. doi: 10.1093/jjco/hyx067. PMID 28582510
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com